CLINICAL TRIAL: NCT00476697
Title: The Effectiveness of UVA1 Irradiation in the Treatment of Skin Conditions With Altered Dermal Matrix: An Open Pilot Study
Brief Title: UVA1 Light for Scleroderma and Similar Conditions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inactivity
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yolanda Rosi Helfrich, Director Program for Clinical Research In Dermatology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Derm 364
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Keloid; Scleroderma; Scars; Granuloma Annulare; Acne Keloidalis Nuchae
Keywords: UVA1; scleroderma; keloids; morphea; light therapy
MeSH Terms: conditions — Keloid; Scleroderma, Diffuse; Cicatrix; Granuloma Annulare; Acne Keloid; Scleroderma, Localized

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UVA1 Irradiation (Experimental): UVA1 irradiaton up to 5 times per week, for up to 16 weeks using German manufactured UVA1 emitting light system. UVA1 dose will be applied with up to 130 J/cm2.
  Interventions: Device: German manufactured UVA1 emitting light system

INTERVENTIONS:
Device: German manufactured UVA1 emitting light system — The dose and scheduling of irradiation is as follows: Up to 130J/cm2 from a UVA1 Sellamed irradiation device with irradiations up to 5 times per week.

SUMMARY:
The purpose of this investigation is to evaluate the effectiveness of high-dose UVA1 irradiation in the treatment of fibrosing conditions of the skin, e.g., keloid (a thick scar from growth of fibrous tissue), scleroderma (deposits of fibrous tissue in the skin) and acne keloidalis nuchae (keloids on the back of the neck or hairline) old burn scars, granuloma annulare or other similar skin conditions. This UVA1 dosing schedule has been used successfully in Germany for various skin diseases, such as the above mentioned scleroderma.

DETAILED DESCRIPTION:
Ultraviolet rays from the sun that reach the earth surface are divided into shorter wavelength, hence high energy, UVB (290-320nm) and longer wavelength, hence low energy UVA (320-400nm). The wavelengths of light that cause sunburn and are associated with skin cancer causation is the high energy UVB. UVA wavelengths can be further divided into relatively shorter wavelength, hence higher energy UVA2 (320-340nm) and longer wavelength, lower energy UVA1 (340-400nm). Phototherapy light boxes used in our clinic for the treatment of psoriasis, atopic dermatitis, and pruritus, as well as those used in tanning salons emit both UVB and UVA wavelengths of light. The advantages of using UVA1 light source in the treatment of skin conditions are 1) lack of skin cancer and sunburn causing rays (UVB) and 2) as a consequence, the ability to treat patients more safely and longer.

Keloid, scleroderma, acne keloidalis nuchae, and burn scars are all characterized by collagenous thickening of the skin resulting in superficial and deep cutaneous sclerosis. Treatments for these disabling conditions are inadequate at present. Recently, in non-controlled studies, UVA1 was shown to induce improvement in patients with scleroderma, granuloma annulare and urticaria pigmentosa (1-3). The mode of action of UVA1 treatment is not completely understood, however, local immuno-modulation appears to be important (4). UVA1 has also been shown to stimulate collagenase activity in a dose dependent manner in the dermis (5,6). We postulate, therefore, that UVA1 in appropriate doses can improve these fibrosing skin conditions safely through collagenase-mediated removal of excess dermal collagen.

Based on the result of this pilot study, a formal controlled clinical investigation is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10-80 years
* Clinical diagnosis of keloid (or hypertrophic scar), scleroderma, acne keloidalis nuchae, old burn scars, granuloma annulare, and other related conditions associated with altered dermal matrix.
* No disease states or physical conditions which would impair evaluation of the test site.
* Willing and able to receive UVA1 as directed in the protocol, make evaluation visits, and follow protocol restrictions.
* Signed, written, witnessed, informed consent form.
* Must live within driving distance of Ann Arbor, Michigan.

Exclusion Criteria:

* History of photosensitivity.
* Pregnant or nursing women.
* Systemic therapy for the fibrosing skin condition within 30 days prior to study enrollment.
* Involved in an investigational study within the previous 4 weeks.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1997-01; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Measurement of plaque thickness, increase in mobility, plaque hardness | 16 weeks

SECONDARY OUTCOMES:
Analysis of collagen levels, mmp induction | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Helfrich, MD, Principal Investigator — University of Michigan hospital
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States